CLINICAL TRIAL: NCT02129439
Title: SB012 for Treatment of Active Ulcerative Colitis: Prospective Multi-centre Randomised Double-blind Placebo-controlled Phase IIa Clinical Trial to Evaluate Efficacy, Pharmacokinetics, Tolerability and Safety of SB012 Enema Administered OD
Brief Title: Efficacy, Pharmacokinetics, Tolerability, Safety of SB012 Intrarectally Applied in Active Ulcerative Colitis Patients
Acronym: SECURE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB012/01/2013
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2017-07

CONDITIONS: Colitis, Ulcerative
Keywords: Antisense oligonucleotide; Colitis Ulcerosa; Ulcerative colitis; Phase II; Transcription factor GATA-3; intrarectal application; proof-of-concept
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB012 (Experimental): SB012 will be available in this clinical trial in a concentration of 7.5 mg/ml hgd40 in 30ml PBS. The maximum daily dose will not exceed 225mg.
  The study will be continued until 18 subjects have completed the four-week treatment phase according to te protocol. 12 of the 18 subjects will receive verum SB012 (in a 2:1 randomization SB012:Placebo)
  Interventions: Drug: SB012
- Placebo (Placebo Comparator): Placebo will be administered with an identical volume of 30ml PBS.
  The study will be continued until 18 subjects have completed the four-week treatment phase according to te protocol. 6 of the 18 subjects will receive placebo (in a 2:1 randomization SB012:Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB012 — The treatment phase lasts 28 consecutive days. The IMP will be administered for the first time at the study site in the morning on Day 1 (IMP administration training by study site staff). The final administration will be performed at the study site in the morning of Day 28. On all other treatment days (Day 2 to Day 27), the IMP will be self-administered by the subject at home.
  SB012 will be available in this clinical trial in a concentration of 7.5mg/ml hgd40 in 30ml PBS (Maximum daily dose: 225mg)
  The IMP is formulated as an enema and will be administered in this clinical trial by the rectal route. The enema is a ready-for-use preparation. No further preparation steps are required.
  No modifications are permitted to the dosing regimen except for premature study discontinuation.
  Other Names: Active drug substance is hgd40
  Arms: SB012
Drug: Placebo — Intervention of placebo-treated subjects does not vary to SB012-treated subjects.
  The treatment phase lasts 28 consecutive days. Placebo will be administered for the first time at the study site in the morning on Day 1 (Administration training by study site staff). The final administration will be performed at the study site in the morning of Day 28. On all other treatment days (Day 2 to Day 27), the IMP/Placebo will be self-administered by the subject at home. Placebo will be administered with a volume of 30ml.
  The IMP/Placebo is formulated as an enema (plastic rectal tube) and will be administered in this clinical trial by the rectal route. The enema is a ready-for-use preparation. No further preparation steps are required.
  Other Names: Active ingredient-free PBS solution
  Arms: Placebo

SUMMARY:
Ulcerative colitis (UC) represents one of the major entities of idiopathic inflammatory bowel diseases which are defined as chronically relapsing inflammations of the gastrointestinal tract not due to specific pathogens. It is characterised by a superficial, continuous mucosal inflammation, which predominantly affects the large intestine. The clinical course is typically marked by periods of asymptomatic remission punctuated by unpredictable recurrent attacks. The symptoms of the patients are marked by persistent diarrhoea with severe faecal urgency and often incontinence, rectal bleeding, abdominal cramping and weight loss.

Uncontrolled activation of mucosal effector T cells has been identified as the main pathogenic mechanism involved in the initiation and perpetuation of intestinal inflammatory reactions.

Patients with moderate UC are initially treated with mesalazine, applied both orally and rectally. If symptoms do not improve, systemic corticosteroids are to be administered. Patients who do not respond to systemic corticosteroids may become eligible for treatment with a calcineurin inhibitor or an anti-tumor necrosis factor (TNF)α antibody. Alternatively, patients may have to undergo major colorectal surgery.

Patients who do not adequately respond to these treatment strategies exhibit serious drawbacks. Colorectal surgery may result in a severely compromised quality of life.

Therefore, patients with moderate or severe UC may significantly benefit from new therapeutic alternatives.

The transcription factor GATA-3 is an interesting target for a novel therapeutic strategy in UC.

GATA-3 is the key regulation factor of Th2-driven immune responses. It is indispensable for the differentiation and activation of Th2 cells, integrates Th2 signals, and induces Th2 cytokine expression. Results of a recent clinical trial in children showed that GATA-3 is involved in the pathogenesis of the acute phase of UC.

The investigational product SB012 contains the DNAzyme hgd40 that targets GATA-3. By cleaving GATA-3 mRNA hgd40 reduces specific cytokine production and thereby reduces key features of mucosal inflammation.

DNAzymes are completely generated by chemical synthesis, not by use of any living organism and are therefore not biological drugs.

This study will evaluate the efficacy, safety, tolerability and pharmacokinetics of the topical formulation SB012 available in a concentration of 7.5mg/ml hgd40 in 30ml PBS once daily as a ready-for-use enema in patients with active UC.

ELIGIBILITY:
Inclusion Criteria:

The trial population consists of adult subjects of both sexes with active ulcerative colitis aged 18 to 75 years.

The main inclusion criteria comprise:

* Fully capable to give informed consent.
* Mentally able to understand the nature, significance, implications and risks of the clinical trial and to follow instructions of the trial staff.
* Written informed consent
* Clinical Mayo Score of ≥3
* Total Mayo Score of ≥6
* Endoscopic Mayo score ≥2 in the sigmoid
* Body mass index ≥18.0 to ≤29.0kg/m2 and body weight ≥50 to ≤100kg
* Negative urine pregnancy test (female subject only)
* Using two methods of contraception

Exclusion Criteria:

* Colectomy and presence of ileal pouch-anal anastomosis or ileorectal anastomosis
* Diagnosis of ulcerative proctitis, fulminant colitis, toxic megacolon, of colitis indeterminata or Crohn's disease
* Ileostoma
* Anti-TNFα treatment with adalimumab, certolizumab, etanercept, golimumab, or infliximab ≤4 weeks prior to screening visit.
* Change in systemic glucocorticoid treatment ≤1 weeks prior to screening visit
* Change in 5-Aminosalicylic Acid (ASA) therapy ≤1 week prior to screening visit
* Start of treatment with an immunosuppressive agent ≤3 months prior to screening visit
* Change in treatment with an immunosuppressive agent ≤4 weeks prior to baseline visit
* Planned concomitant therapeutic administration of suppositories or foams or enema other than the IMP.
* Impaired blood coagulation (Quick value <50% and/or partial thromboplastin time (PTT) >55sec and/or platelet count <50.000/μl.)
* Signs of renal insufficiency
* Signs of hepatic insufficiency.
* Current treatment with drugs of high hepatotoxic potential.
* Evidence of recent alcohol abuse.
* Acute or chronic heart failure with NYHA functional class III or IV.
* Known active tuberculosis.
* Known acute serious infections or sepsis.
* Known current malignant disease.
* Positive blood test against HBs antigen, anti-HBc antibodies, anti-HCV antibodies or anti-HIV-1/2 antibodies.
* Known opportunistic infections including invasive fungal infections.
* Known hypersensitivity to the IMP or any of their formulation ingredients.
* Any condition that is thought to reduce the compliance to cooperate with the trial procedures.
* Employee of the department of the investigator, of the Center for Clinical Studies (CCS) or of the sponsor.
* Prior participation in this clinical trial.
* Participation in an interventional clinical trial within the last three months (six months in case of a biological IMP) or be under the exclusion period from another clinical trial.
* Known or planned absence that may collide with the clinical trial visit schedule.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Efficacy: Total Mayo score (4 weeks comparison) | Baseline (Visit 2) to day 28 (Visit 7) (28 days)
  Change in Total Mayo score after 4 weeks of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
  The Total Mayo score is a 13-point ordinal scale for the assessment of concurrent severity of ulcerative colitis. It comprises four components: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment of disease severity. Each component has four grades ranging from 0 to 3. The Total Mayo score ranges from 0 to 12, with 12 representing the most severe disease.

SECONDARY OUTCOMES:
Efficacy: Total Mayo score (8 weeks comparison) | Baseline (Visit 2) to End-of-Study Visit10 (56 days)
  Change in Total Mayo score 8 weeks after start of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
Efficacy: Endoscopic Mayo score (4 and 8 weeks comparison) | Baseline (Visit 2) to Visit 7 and Visit 10 (28 and 56 days)
  Change in Endoscopic Mayo score 4 and 8 weeks after start of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
  The Endoscopic Mayo score represents a subscore of the Total Mayo score and consists of the endoscopic findings. It ranges from 0 to 3.
  Normal or inactive disease 0 Mild disease (erythema, decreased vascular pattern, mild friability) 1 Moderate disease (marked erythema, absent vascular pattern, friability, erosions) 2 Severe disease (spontaneous bleeding, ulceration) 3
Efficacy/Pharmacodynamics: Glucocorticoid consumption | Baseline (Visit 2) to day 56 End of Study Visit 10 (56 days)
  Change in systemic glucocorticoid consumption (measured as Defined Daily Dose) 8 weeks after start of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
Safety: Treatment Emergent Adverse Events (AE) and Serious Adverse Events (SAE) | Visit 1 (Screening) to Visit 10 (End of Study - 56 days) or Visit X (Early Study Termination)
  Number of treatment-emergent AEs and SAEs in the active treatment group (SB012) versus placebo in patient´s overall study period.

OTHER OUTCOMES:
Pharmacokinetic (PK) analysis | First treatment Day 1/day 2 (Visit 3/4) to Last treatment day 28/29 (Visit 7/8)
  In subjects with hgd40 plasma levels equal to or above "lower limit of quantification" (LLOQ): mean hgd40 plasma concentrations per time point.
  Blood sampling for PK analysis prior to IMP administration and 1, 2, 4, 6 and 24 hours after IMP administration with a time window of ±2min for the 1 and 2 hour time point, of ±5min for the 4 and 6 hour time points and a time window of ±1 h for the 24 hour time point.
Exploratory analysis: Systemic biomarker plasma levels | Day 1 (Visit 3) to Day 28 or Day 56 (V7 or V10)
  To evaluate the effects of SB012 enema on disease activity assessed by histology of, and biomarker expression in, biopsies from affected colonic tissue and on systemic biomarker expression in the blood.
Exploratory analysis: Systemic biomarker plasma levels | Day 1 (Visit 3) to Day 28 or Day 56 (V7 or V10)
  Change in GATA-3 mRNA expression 4 and 8 weeks after start of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
Exploratory analysis: Riley Score | Day 1 (Visit 3) to Day 28 or Day 56 (V7 or V10)
  Change in Riley score 4 and 8 weeks after start of treatment compared to baseline value in the active treatment group (SB012) versus placebo.
  The Riley score is a 19-point ordinal scale for the quantification of inflammatory activity in tissue affected by ulcerative colitis based on the following six histological criteria :
  * Acute inflammatory cell infiltrates (polymorphonuclear).
  * Crypt abscesses.
  * Mucin depletion.
  * Surface epithelial integrity.
  * Chronic inflammatory cell infiltrate.
  * Crypt architectural irregularities.
  Each criterion has a grade ranging from 0 to 3, with 18 representing the most severe state of inflammation:
  Score Inflammation
  * None 0
  * Mild 1
  * Moderate 2
  * Severe 3

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, Prof. Dr., Principal Investigator — Department of Medicine 1 - Gastroenterology, Pneumology and Endocrinology, University Clinic Erlangen, Germany
Locations (3):
- Germany (3):
  - Braunschweig Municipal Hospital - Medical Clinic 1, Braunschweig
  - Department of Medicine 1 - Gastroenterology, Pneumology and Endocrinology, University Clinic Erlangen, Germany, Erlangen
  - Asklepios West Hospital Hamburg - Division Gastroenterology, Hamburg